CLINICAL TRIAL: NCT03086772
Title: Effects of Tai Chi on Multisite Pain and Brain Functions in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tongjian You, Associate Professor, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AG043883 (NIH); R21AG043883 (NIH)
Record Dates: First submitted 2015-06-04; First posted 2017-03-22 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Experimental): Individuals in the Tai Chi intervention group participated in a 12-week Tai Chi program.
  Interventions: Behavioral: Tai Chi
- Light Exercise (Active Comparator): Individuals in the exercise control group performed a 12-week light exercise program.
  Interventions: Behavioral: Light Exercise

INTERVENTIONS:
Behavioral: Tai Chi — Individuals in the Tai Chi intervention group will participate in a 12-week Tai Chi program (one hour per class, two classes per week, plus home practice for 12 weeks) led by an experienced Tai Chi Instructor, assisted by an undergraduate research assistant.
  Arms: Tai Chi
Behavioral: Light Exercise — Individuals in the exercise control group will meet for a twice weekly class involving walking, weight training, stretching and health education (one hour per class, two classes per week for 12 weeks, taught by a trained graduate research assistant, assisted by an undergraduate research assistant.
  Arms: Light Exercise

SUMMARY:
The main purpose of this randomized controlled trial was to assess the feasibility and acceptability of a 12-week Tai Chi program for community-dwelling older adults with chronic multisite pain and a history of falling. In addition, the investigators examined the effects of Tai Chi on pain characteristics, cognition, physical function, gait mobility, levels of pain-related biomarkers, fear of falling and rate of falls in these older adults.

DETAILED DESCRIPTION:
Older adults aged ≥65 years with multisite pain who reported falling in the past year or current use of an assistive device were recruited from Boston area communities. Participants were randomized to either a Tai Chi (N=28) or a light physical exercise (N=26) program, offered twice weekly for 12 weeks. The primary outcomes were feasibility and acceptability of the 12-week Tai Chi/light exercise program. Secondary outcomes included pain characteristics (pain severity and pain interference), cognition (attention and executive function), physical function (walking speed, strength, and balance), gait mobility (singe-task and dual-task gait), levels of pain-related markers (C-reactive protein, interleukin 6, tumor necrosis factor alpha, and beta endorphin), fear of falling, and rate of falls.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years and older
* Multisite (2 or more sites) musculoskeletal pain
* At least one fall in the past year, or currently on an assistive device
* A sedentary lifestyle
* Be able to walk 20-feet without personal assistance
* Be able to communicate in English.

Exclusion Criteria:

* Regular Tai Chi practice
* Unstable cardiac disease
* Stroke
* Rheumatoid arthritis
* Degenerative neuromuscular disease
* Parkinson's disease
* Terminal disease
* Dementing illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the 12-week Tai Chi program | Over the 12-week intervention period
  Feasibility and acceptability were evaluated by adherence, attendance, optimal program components, and safety.

SECONDARY OUTCOMES:
Pain characteristics | Before and after the 12-week intervention period
  Pain severity and interference were evaluated by using the Brief Pain Inventory (BPI) questionnaire.
Cognition | Before and after the 12-week intervention period
  Attention was evaluated by using the Test of Everyday Attention (TEA) questionnaire. Executive function was evaluated by using the Trailmaking A and B tests questionnaire.
Physical function | Before and after the 12-week intervention period
  Physical function was measured by using the Short Physical Performance Battery (SPPB)
Gait mobility | Before and after the 12-week intervention period
  Single-task and dual-task gait function was determined by using the PKMAS software and Zeno walkway.
Pain-related biomarkers | Before and after the 12-week intervention period
  Levels of inflammatory markers and beta endorphin were determined by using biochemistry assays.
Fear of falling | Before and after the 12-week intervention period
  Fear of falling was measured using the Tinetti Falls Effi- cacy Scale.
Rate of falls | Over the 12-week intervention and 6 months following the intervention
  Rate of falls were recorded by using monthly fall calendars.

CONTACTS AND LOCATIONS:
Overall Officials: Tongjian You, PhD, Principal Investigator — University of Massachusetts, Boston; Suzanne Leveille, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- University of Massachusetts, Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] You T, Ogawa EF, Thapa S, Cai Y, Zhang H, Nagae S, Yeh GY, Wayne PM, Shi L, Leveille SG. Tai Chi for older adults with chronic multisite pain: a randomized controlled pilot study. Aging Clin Exp Res. 2018 Nov;30(11):1335-1343. doi: 10.1007/s40520-018-0922-0. Epub 2018 Mar 6. PMID 29512041